CLINICAL TRIAL: NCT02603523
Title: Effects of Senior Dance on Risk Factors for Falls in Older Adults: A Randomized Controlled Trial
Brief Title: Effects of Senior Dance on Risk Factors for Falls
Acronym: DanSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Federal University of Minas Gerais (Other); Universidade Cidade de Sao Paulo (Other); University of Sydney (Other); The George Institute (Other)
Responsible Party: Principal Investigator, Marcia Rodrigues Costa Franco, Dr, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/07704-9
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Accidental Falls
Keywords: accidental falls; older people; dance; randomized controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Senior Dance (Experimental): The intervention group will attend a single educational class on fall risk factors and prevention, and will participate in a 12-week, twice-weekly group-based program of Senior Dance. Each dance class will last for an hour, and the number of participants per class will range from 10 to 15. Senior Dance-certified instructors will lead the classes. The Senior Dance classes consist of different choreographies, which include rhythmic and simple movements with rhythmic folk songs. During the classes, participants can practice the movements sitting or standing, quickly or slowly, in circles, individually, in pairs or in small groups.
  Interventions: Behavioral: Senior Dance
- Control group (No Intervention): Participants in the control group will attend the same educational class on fall risk factors and prevention that intervention group participants will receive, and will be instructed not to take part in any regular exercise programs such as supervised group exercise, Tai Chi, Yoga, or any dance activity during the study period. At the end of the study, they will be offered Senior Dance classes, twice a week, during 12 weeks.

INTERVENTIONS:
Behavioral: Senior Dance — The Senior Dance classes consist of different choreographies, which include rhythmic and simple movements with rhythmic folk songs. During the classes, participants can practice the movements sitting or standing, quickly or slowly, in circles, individually, in pairs or in small groups. The concentration required to learn the choreographies challenges balance, motor coordination and cognitive function.
  Arms: Senior Dance

SUMMARY:
The efficacy of exercise programs to prevent falls among older people is well documented in the literature. However, older people's adherence to these exercise programs has been reported to be suboptimal, varying between 21% and 74%. In addition, about 45% of people aged over 60 years do not meet the minimum recommended level of physical activity. In this context, dance is a promising alternative to traditional exercise programs, as it can positively influence important risk factors for falls, such as sedentary lifestyle, balance impairments and muscle weakness. Nevertheless, a recent systematic review conducted in this area show that the lack of randomized clinical trials as well as the low methodological quality of existing studies do not allow to reach definitive conclusions on the real effects of dance on risk factors for falls. A type of dance that is becoming popular among the older population in Brazil is the Senior Dance. Senior Dance classes consist of different choreographies, which include rhythmic and simple movements with rhythmic folk songs. The concentration required to learn the choreographies challenges balance, motor coordination and cognitive function. Thus the present study is a randomized clinical trial aiming to investigate the Senior Dance effect on balance, mobility and cognitive function, compared with a control group, among older people living in the community. A total of 82 subjects will be randomly allocated into two groups. The intervention group will participate in a 12-week, twice-weekly group-based program of Senior Dance, while the control will be encouraged to maintain their current routine activities. Outcomes measures (balance, mobility and cognitive function) will be evaluated before and after the intervention by an assessor blinded to group allocation. The results of this study will assist health practitioners when prescribing intervention for the older population.

ELIGIBILITY:
Inclusion criteria:

* Community-dwelling aged 60 years or over
* Cognitively intact (defined as a minimum score of 24 points on the Mini Mental Status Examination).

Exclusion criteria:

* Previous stroke with severe neurological impairment
* Progressive neurological disease
* Severe visual deficiency, dizziness or vertigo for less than 3 months
* Inability to maintain a standing position, even with the use of a walking aid or other device
* Any illness that the physician considers as an exercise contra-indication (e.g. uncontrolled angina, acute coronary disease).
* Participants who are currently participating in regular exercise programs including strength training and balance challenge, such as supervised group exercise, Tai Chi, Yoga, or any dance activity.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Single-leg stance with eyes closed | 12 weeks after randomization

SECONDARY OUTCOMES:
Short Physical Performance Battery | 12 weeks after randomization
Falls Efficacy Scale - International (FES-I) | 12 weeks after randomization
Trail Making Test (TMT) | 12 weeks after randomization
The Montreal Cognitive Assessment (MOCA): | 12 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Marcia R Franco, PhD, Principal Investigator — Departamento de Fisioterapia, Faculdade de Ciências e Tecnologia, UNESP - Universidade Estadual Paulista, Presidente Prudente, São Paulo, Brasil; Carlos Marcelo Pastre, PhD, Study Director — Departamento de Fisioterapia, Faculdade de Ciências e Tecnologia, UNESP - Universidade Estadual Paulista, Presidente Prudente, São Paulo, Brasil
Locations (1):
- UNESP, Presidente Prudente, São Paulo, Brazil

REFERENCES:
- [Background] Fernandez-Arguelles EL, Rodriguez-Mansilla J, Antunez LE, Garrido-Ardila EM, Munoz RP. Effects of dancing on the risk of falling related factors of healthy older adults: a systematic review. Arch Gerontol Geriatr. 2015 Jan-Feb;60(1):1-8. doi: 10.1016/j.archger.2014.10.003. Epub 2014 Nov 6. PMID 25456888
- [Derived] Franco MR, Sherrington C, Tiedemann A, Pereira LS, Perracini MR, Faria CSG, Negrao-Filho RF, Pinto RZ, Pastre CM. Effect of Senior Dance (DanSE) on Fall Risk Factors in Older Adults: A Randomized Controlled Trial. Phys Ther. 2020 Apr 17;100(4):600-608. doi: 10.1093/ptj/pzz187. PMID 31899491
- [Derived] Franco MR, Sherrington C, Tiedemann A, Pereira LS, Perracini MR, Faria CR, Pinto RZ, Pastre CM. Effectiveness of Senior Dance on risk factors for falls in older adults (DanSE): a study protocol for a randomised controlled trial. BMJ Open. 2016 Dec 30;6(12):e013995. doi: 10.1136/bmjopen-2016-013995. PMID 28039296